CLINICAL TRIAL: NCT06538441
Title: Dynamic Pattern of Etiology, Immunoinflammatory Factors and Their Association With Prognosis of Severe Pneumonia: a Longitudinal Observational Study
Brief Title: Dynamic Pattern of Etiology, Immunoinflammatory Factors and Their Association With Prognosis of Severe Pneumonia
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai General Hospital, China (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Mei Kang, Principal Investigator, Shanghai General Hospital, China
Other Study IDs: 2024023
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Severe Pneumonia
Keywords: Pneumonia; Etiology; Inflammatory factor; Disease Progression; Prognosis
MeSH Terms: conditions — Pneumonia; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe pneumonia: Severe pneumonia patients will be continuously recruited in ICU department in Shanghai General Hospital (n=450) and RICU in the First Affiliated Hospital of Chongqing Medical University (n=150) during June 1, 2022 to April 28, 2024.
  Severe pneumonia was defined as meeting either one major criteria (septic shock with need of vasopressors or respiratory failure requiring mechanical ventilation) or three minor (laboratory and physiologic markers such as uremia or hypothermia) criteria according to the ATS/IDSA major criteria.

SUMMARY:
The goal of this longitudinal observational study is to investigate the pathogen spectrum composition of severe pneumonia (SP) in different disease stages and to study the changes of immune inflammatory factors in patients with SP in different course of disease during and after the COVID-19 pandemic. The main questions it aims to answer is:

What is the pathogenic profile of SP patient admitted in intensive care unit (ICU) during and after COVID-19 pandemic? What is the dynamic pattern of etiology and immunoinflammatory factors of SP progression during the period in ICU? Are those indexes mentioned above associated with the prognosis of SP?

DETAILED DESCRIPTION:
This is a multi-center, longitudinal, observational study.

Participants

SP patients will be continuously recruited in ICU department in Shanghai General Hospital and respiratory-specific ICU (RICU) department in the First Affiliated Hospital of Chongqing Medical University during June 1, 2022 to December 31, 2024.

The investigators applied the AmericanThoracic Society(ATS)/Infectious Diseases Society of America (IDSA) major criteria to a cohort of patients hospitalized in two tertiary hospitals with severe pneumonia in order to describe its epidemiology, microbiology, and outcomes.

Assessment of disease progression

1. Shock: Definition: A systemic pathological process in which the effective circulating blood volume is reduced due to various reasons and the tissue microcirculation perfusion is seriously insufficient, resulting in cell damage and serious dysfunction of function and metabolism of important organs. Overall arterial pressure decline: systolic blood pressure less than 90mmHg or mean arterial pressure (MAP) less than 70mmHg, accompanied by tachycardia. Clinical signs of hypoperfusion: skin damp cold with vasoconstriction and cyanosis; Kidney urine volume is less than 0.5ml/kg/h; The nervous system includes changes in mind (dullness of reaction, loss of orientation and confusion). Hyperlactacidemia: greater than 2mmol/L.
2. Invasive mechanical ventilation: (1) Definition: Support of ventilation and improvement of oxygenation by inserting an intubation tube into the trachea and delivering warm, fully oxygenated, and moist gases to the airways and lungs at pressures above atmospheric pressure. (2) Classification: invasive ventilator-assisted ventilation under tracheal intubation, invasive ventilator-assisted ventilation under tracheal incision.
3. High fever: body temperature (armpit temperature) exceeds 39 ° C. (Note: High fever is generally defined at 38.5℃ in clinical practice.)
4. The above symptoms persist: shock for more than 3 days, high fever for more than 3 days, mechanical ventilation for more than 1 week.

Indicators

1. Sociodemographic indexes: sex, age, personal history
2. Clinical indicators: clinical diagnosis, past history, present history, treatment history, laboratory examination, clinical prognosis
3. Laboratory examination : culture, species of infectious agent, antibiotic susceptibility test Microbiological etiological identification methods include: ① oral and pharyngeal swabs: polymerase chain reaction (PCR) for COVID-19 nucleic acid; ② Nasopharyngeal swab: PCR for influenza A virus nucleic acid; ③ Rectal swab: Macconkey plate + drug-sensitive paper was used to detect the presence of carbapenem-resistant gram-negative bacillus, and loop-mediated isothermal amplification was used to identify the presence of IPM, VIM, NDM, KPC, OXA and other resistance genes. ④ Smear: Various specimens are diluted and stained to observe whether there are bacteria and fungi and their morphology; ⑤ Culture: microbial culture of various specimens, and drug sensitivity test to determine drug resistance; ⑥ Quick test: Rapid detection of infectious diseases, including 17 bacteria and 7 fungi; ⑦ Immunofluorescence staining: Use fluorescein to label fungal cell wall, observe fungal morphology under fluorescence microscope for qualitative detection; ⑧ Next generation sequencing (NGS).

Other laboratory tests: Blood routine (white blood cell count, neutrophil count, lymphocyte count and neutrophil-to-lymphocyte ratio (NLR), C-reactive protein (CRP), procalcitonin (PCT)).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Clinical diagnosed of severe pneumonia (case definition: adults according to "Diagnosis and Treatment of Adults with Community-acquired Pneumonia"-- An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America, 2019)
* Have at least one microbiological test result

Exclusion Criteria:

* No data of clinical prognosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe pneumonia patients admitted in ICU department in Shanghai General Hospital and respiratory-specific ICU department in the First Affiliated Hospital of Chongqing Medical University during June 1, 2022 to April 28, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | up to 3 months
  Number of Participants with fatal outcomes out of all participants

SECONDARY OUTCOMES:
length of stay in ICU | through study completion, an average of 38 days
  Number of days since admitted to ICU for each patient
duration of mechanical ventilation | through study completion, an average of 25 days
  Number of days of mechanical ventilation treatment for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Mei Kang, MPH, Principal Investigator — Clinical Research Center, Shanghai General Hospital
Locations (1):
- Mei Kang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used in this study are available upon request to the principle investigator.

REFERENCES:
- [Background] Drigot ZG, Clark SE. Insights into the role of the respiratory tract microbiome in defense against bacterial pneumonia. Curr Opin Microbiol. 2024 Feb;77:102428. doi: 10.1016/j.mib.2024.102428. Epub 2024 Jan 25. PMID 38277901
- [Background] Azoulay E, Russell L, Van de Louw A, Metaxa V, Bauer P, Povoa P, Montero JG, Loeches IM, Mehta S, Puxty K, Schellongowski P, Rello J, Mokart D, Lemiale V, Mirouse A; Nine-i Investigators. Diagnosis of severe respiratory infections in immunocompromised patients. Intensive Care Med. 2020 Feb;46(2):298-314. doi: 10.1007/s00134-019-05906-5. Epub 2020 Feb 7. PMID 32034433
- [Background] Natalini JG, Singh S, Segal LN. The dynamic lung microbiome in health and disease. Nat Rev Microbiol. 2023 Apr;21(4):222-235. doi: 10.1038/s41579-022-00821-x. Epub 2022 Nov 16. PMID 36385637
- [Background] Shi Y, Huang Y, Zhang TT, Cao B, Wang H, Zhuo C, Ye F, Su X, Fan H, Xu JF, Zhang J, Lai GX, She DY, Zhang XY, He B, He LX, Liu YN, Qu JM. Chinese guidelines for the diagnosis and treatment of hospital-acquired pneumonia and ventilator-associated pneumonia in adults (2018 Edition). J Thorac Dis. 2019 Jun;11(6):2581-2616. doi: 10.21037/jtd.2019.06.09. No abstract available. PMID 31372297
- [Background] Simon L, Gauvin F, Amre DK, Saint-Louis P, Lacroix J. Serum procalcitonin and C-reactive protein levels as markers of bacterial infection: a systematic review and meta-analysis. Clin Infect Dis. 2004 Jul 15;39(2):206-17. doi: 10.1086/421997. Epub 2004 Jul 2. PMID 15307030
- [Background] Xie Y, Du J, Jin W, Teng X, Cheng R, Huang P, Xie H, Zhou Z, Tian R, Wang R, Feng T. Next generation sequencing for diagnosis of severe pneumonia: China, 2010-2018. J Infect. 2019 Feb;78(2):158-169. doi: 10.1016/j.jinf.2018.09.004. Epub 2018 Sep 18. No abstract available. PMID 30237069
- [Background] Kelly BJ, Imai I, Bittinger K, Laughlin A, Fuchs BD, Bushman FD, Collman RG. Composition and dynamics of the respiratory tract microbiome in intubated patients. Microbiome. 2016 Feb 11;4:7. doi: 10.1186/s40168-016-0151-8. PMID 26865050
- [Background] Yang L, Haidar G, Zia H, Nettles R, Qin S, Wang X, Shah F, Rapport SF, Charalampous T, Methe B, Fitch A, Morris A, McVerry BJ, O'Grady J, Kitsios GD. Metagenomic identification of severe pneumonia pathogens in mechanically-ventilated patients: a feasibility and clinical validity study. Respir Res. 2019 Nov 27;20(1):265. doi: 10.1186/s12931-019-1218-4. PMID 31775777
- [Background] Huang WC, Wu MF, Huang CC, Liu SY, Chen HC, Chen YY, Hsu JY, Huang CC. Dynamics of the lung microbiome in intensive care patients with chronic obstructive pulmonary disease and community-acquired pneumonia. Sci Rep. 2020 Jul 6;10(1):11046. doi: 10.1038/s41598-020-68100-4. PMID 32632240
- [Background] Shi N, Huang C, Zhang Q, Shi C, Liu F, Song F, Hou Q, Shen J, Shan F, Su X, Liu C, Zhang Z, Shi L, Shi Y. Longitudinal trajectories of pneumonia lesions and lymphocyte counts associated with disease severity among convalescent COVID-19 patients: a group-based multi-trajectory analysis. BMC Pulm Med. 2021 Jul 13;21(1):233. doi: 10.1186/s12890-021-01592-6. PMID 34256743
- [Background] Lin MJ, Rachleff VM, Xie H, Shrestha L, Lieberman NAP, Peddu V, Addetia A, Casto AM, Breit N, Mathias PC, Huang ML, Jerome KR, Greninger AL, Roychoudhury P. Host-pathogen dynamics in longitudinal clinical specimens from patients with COVID-19. Sci Rep. 2022 Apr 7;12(1):5856. doi: 10.1038/s41598-022-09752-2. PMID 35393464
- [Background] File TM Jr, Ramirez JA. Community-Acquired Pneumonia. N Engl J Med. 2023 Aug 17;389(7):632-641. doi: 10.1056/NEJMcp2303286. No abstract available. PMID 37585629
- [Background] Xie L, Luo G, Yang Z, Wu WC, Chen J, Ren Y, Zeng Z, Ye G, Pan Y, Zhao WJ, Chen YQ, Hou W, Sun Y, Guo D, Yang Z, Li J, Holmes EC, Li Y, Chen L, Shi M. The clinical outcome of COVID-19 is strongly associated with microbiome dynamics in the upper respiratory tract. J Infect. 2024 Mar;88(3):106118. doi: 10.1016/j.jinf.2024.01.017. Epub 2024 Feb 10. PMID 38342382
- [Background] Perez-Cobas AE, Baquero F, de Pablo R, Soriano MC, Coque TM. Altered Ecology of the Respiratory Tract Microbiome and Nosocomial Pneumonia. Front Microbiol. 2022 Feb 10;12:709421. doi: 10.3389/fmicb.2021.709421. eCollection 2021. PMID 35222291